CLINICAL TRIAL: NCT03478345
Title: Taking Action to Thrive - A Healthy Lifestyle Intervention Pilot Study
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Kimberly Robien, Associate Professor, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111739
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Overweight, Obesity and Other Hyperalimentation
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THRIVE Study (Experimental)
  Interventions: Behavioral: endocrine disruptor chemical reduction intervention

INTERVENTIONS:
Behavioral: endocrine disruptor chemical reduction intervention — Participants will take part in a 4-week intervention consisting of a modified (shortened) version of the Diabetes Prevention Program diet and physical activity group education program, with instructions to reduce endocrine disruptor chemical exposure through changes in food handling and personal care products.

SUMMARY:
There have been some preliminary studies, primarily in animals, that suggest that exposure to some of the chemicals in our everyday environment, such as the chemicals found in plastics, may cause weight gain. It is not clear whether this also happens in humans, or whether decreasing exposure to these chemicals can improve success with weight loss when people adopt healthy lifestyle changes.

The THRIVE Study is a 4-week group healthy lifestyle education program that is designed to determine whether:

* changes in dietary habits and the types of personal care products used can decrease a person's exposure to chemicals in our environment that have been suggested to cause weight gain
* whether any measurable changes in body composition (fat tissue vs. lean tissue) can be seen as a result of participating in the healthy lifestyle program.

DETAILED DESCRIPTION:
Emerging evidence from in vitro and animal models suggests that exposure to endocrine disrupting chemicals (EDC), or industrial chemicals that alter hormonal action, may contribute to the development of obesity. Phthalates, a class of industrial chemicals commonly found in personal care products and food packaging, warrant study since they are widely detected in the general US population, including reproductive aged-women, and exposures during adulthood are associated with an increased risk of obesity. However, the majority of the evidence supporting this hypothesis to date has come from cross-sectional rather than prospective, longitudinal data. Thus, a causal relationship between EDC exposure and the development of obesity has not been conclusively established.

Currently, 60.3% (95% CI: 54.2-66.0) of younger adult Americans (aged 20 - 39) are thought to be overweight or obese (BMI ≥25), which increases the risk of chronic diseases such as diabetes, cardiovascular disease and cancer. While excess calorie consumption and lack of physical activity are primary contributors to overweight and obesity, factors other than diet and physical activity may also contribute to alterations in energy balance over time. The general public is becoming increasingly concerned about the potential health risks associated with EDC exposures, including effects on body composition.

The THRIVE Study is designed to evaluate the effect of many different EDCs on body composition changes. The study will focus initially on exposures to the phthalate class of EDCs, but data will be collected in a way that will allow investigators to evaluate the effect of many different EDCs on body composition changes.

Phthalates are a class of high-production-volume industrial chemicals that are ubiquitously used in commerce. Most phthalates, such as DEHP, are used as plasticizers to impart flexibility in polyvinyl chloride (PVC) materials such as food packaging, flooring, and medical devices. In recent years, other phthalates, including diisononyl phthalate (DiNP), have been replacing DEHP in these applications due, in part, to legislation limiting the use of DEHP in certain applications such as children's toys. Phthalates can leach, migrate, or off-gas from products over time and enter the human body through the air we breathe, the food we eat, and the personal care products that we use on our bodies. Consequently, human exposure to phthalates is widespread.

Phthalates enter foods through contact with plastics (e.g. tubing, conveyor belts or plastic gloves made with PVC plastics) or recycled paper/cardboard food containers. Phthalates are more likely to leach into liquids and non-polar solvents such as fats and oils, and thus are most commonly found in foods high in animal fats such as dairy products and meat. Low-molecular weight phthalates, such as DEP, di-n-butyl phthalate (DnBP) and DiBP, are commonly found in fragranced personal care products such as perfumes, deodorants, soaps, shampoos, and other hair products (e.g. hair sprays, gels, mousses). They can also be found in time release medications and supplements. Intervention studies suggest that addressing sources of exposure can lower human exposure to phthalates. In a study of 20 individuals, a 3-day dietary intervention of "fresh foods" (no canned food or foods wrapped in plastic) resulted in an average reduction in DEHP metabolites of 53-56%. Similarly, a study of 100 Latina girls found that a 3-day intervention with phthalate free personal care products resulted in a 27.4% reduction in DEP metabolite (mono-ethyl phthalate) levels.

If phthalate exposures are ultimately found to be associated with body composition changes in young adults, it could be possible to decrease the risk of these body composition changes by modifying food selection, preparation and storage techniques, and changing use of personal care products in addition to traditional diet and physical activity interventions. This, in turn, could have significant impacts on obesity and chronic disease risk in the US.

While a few studies have indicated that dietary modification and changes in personal care products use can individually lower urinary phthalate levels, this study will be the first to combine both a dietary and personal care product intervention. In a study of 20 individuals, a 3-day dietary intervention of "fresh foods" (no canned food or foods wrapped in plastic) resulted in an average reduction in DEHP metabolites of 53-56%. Similarly, a study of 100 Latina girls found that a 3-day intervention with phthalate free personal care products resulted in a 27.4% reduction in DEP metabolite (mono-ethyl phthalate) levels. The hypothesis of this study is that an intervention that addresses both dietary and personal care product phthalate exposures can result in an even greater decrease in urinary phthalate metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. female
2. BMI >25 kg/m2
3. willingness to participate in the 4-week long study
4. English speaking
5. capable of giving informed consent.

Exclusion Criteria:

1. males
2. current smoker, or having quit smoking within the past 6 months
3. currently or recently (past 6 months) pregnant or lactating, or planning to become pregnant in the next year
4. engaging in >150 minutes exercise/week
5. weight loss of ≥5 pounds over the past 6 months
6. post-menopausal
7. pre-existing chronic diseases
8. use of medications known to alter body composition such as hormone replacements, oral contraceptives, and steroids
9. homeless persons, or individuals who have active drug/alcohol dependence or abuse history
10. Non-English speaking

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Because of potential hormonal influences on body composition, eligibility criteria for this study requires being biologically female.
Enrollment: 13 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in urinary endocrine disrupting chemical levels (especially phthalates) | Six weeks
  Difference between urinary endocrine disrupting chemical levels from urine collected at the baseline study visit and urine collected at the final study visit.
Changes in body composition (weight and visceral adipose tissue volume) | Six weeks
  Difference between body weight and visceral adipose tissue volume (measured by dual x-ray absorptiometry) from baseline to final study visit.

SECONDARY OUTCOMES:
Correlation between dietary patterns and urinary endocrine disrupting chemical levels | baseline
  Participants will complete three-day food records and urine specimen collections between the baseline study visit and the first group education session. Statistical testing (factor analysis) will be used to determine dietary patterns (e.g. diets high in processed foods or high in fat) that are associated with higher levels of urinary endocrine disrupting chemicals.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Robien, PhD, RD, Principal Investigator — Department of Exercise and Nutrition Sciences, Milken Institute School of Public Health, George Washington University
Locations (1):
- Milken Institute School of Public Health, George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Will not share data until study is complete and all data deidentified